CLINICAL TRIAL: NCT04934072
Title: A Double-blind, Randomized, Multicenter, Multiple-dose, 2-arm, Parallel-group Study to Evaluate Efficacy, Pharmacodynamics, Safety, and Immunogenicity of FKS518 - Proposed Biosimilar to Denosumab With Prolia® in Postmenopausal Women With Osteoporosis (LUMIADE-3 Study)
Brief Title: A Study to Evaluate the Efficacy, Pharmacodynamics, Safety, and Immunogenicity of FKS518 in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FKS518-002; 2020-004422-31 (EudraCT Number)
Record Dates: First submitted 2021-06-03; First posted 2021-06-22 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal Osteoporosis; FKS518; Denosumab; US-licensed Prolia
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — QL1206; Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FKS518 (Experimental): FKS518 was administered on Day 1, and then every 26 weeks (6 months), i.e., Week 26 and Week 52, at a dose of 60 mg for a total of 3 administrations.
  Interventions: Drug: FKS518
- US-Prolia (Active Comparator): US-Prolia was administered on Day 1, and then every 26 weeks (6 months), i.e., Week 26 and Week 52, at a dose of 60 mg for a total of 3 administrations.
  Interventions: Drug: US-licensed Prolia (Amgen)

INTERVENTIONS:
Drug: FKS518 — subcutaneously by single-use prefilled syringe (PFS)
  Other Names: Denosumab biosimilar
  Arms: FKS518
Drug: US-licensed Prolia (Amgen) — subcutaneously by single-use PFS
  Other Names: Denosumab
  Arms: US-Prolia

SUMMARY:
The primary objective of this study is to demonstrate equivalent efficacy of the proposed biosimilar denosumab FKS518 to US-licensed Prolia in women with postmenopausal osteoporosis (PMO).

ELIGIBILITY:
Inclusion Criteria

1. Female ≥55 to ≤85 years of age, inclusive, at screening.
2. Have a body mass index (BMI) ≥18 to ≤32 kg/m^2.
3. Participant should have confirmed postmenopausal status, defined as age-related or early/premature amenorrhea ≥12 consecutive months and increased follicle-stimulating hormone (FSH) >40 mIU/mL at screening; or surgical menopause (bilateral oophorectomy with or without hysterectomy) ≥12 months prior to screening.
4. Absolute bone mineral density (BMD) consistent with T-score ≤-2.5 and ≥-4.0 at the lumbar spine as measured by dual energy x-ray absorptiometry (DXA) as per central assessment.
5. At least 2 vertebrae in the lumbar vertebrae 1 to lumbar vertebrae 4 (L1-L4) region and at least 1 hip joint are evaluable by DXA.
6. Clinically acceptable physical examinations and laboratory tests and no history or evidence of any clinically significant concomitant medical disorder that, in the opinion of the Investigator, would pose a risk to participant safety or interfere with study evaluations or procedures.
7. Written informed consent including accepting a separate Information Sheet containing important information about COVID-19 and its general risks for participants participating in the clinical trial.

Exclusion Criteria:

Disease-related

1. History and/or presence of 1 severe or >2 moderate vertebral fractures or hip fracture confirmed by x-ray.
2. Presence of active healing fracture at screening.
3. History and/or presence of bone-related disorders, such as but not limited to Paget's disease, osteomalacia, hyperparathyroidism (or parathyroid disorders), or renal osteodystrophy.
4. Osteonecrosis of the jaw (ONJ) or risk factors for ONJ such as invasive dental procedures (eg, tooth extraction, dental implants, or oral surgery in the past 6 months), poor oral hygiene, periodontal, and/or pre-existing dental disease as assessed by the Investigator.
5. Evidence of hypocalcemia (albumin-adjusted serum calcium <2.13 mmol/L or <8.5 mg/dL) or hypercalcemia (albumin-adjusted serum calcium >2.6 mmol/L or >10.5 mg/dL) as assessed by the central laboratory at screening.
6. Vitamin D deficiency (25-hydroxy vitamin D levels <12 ng/mL) as assessed by central laboratory at screening (retest is allowed once).
7. Known intolerance to calcium or vitamin D supplements.

   Other Medical Conditions
8. Known or suspected clinically relevant drug hypersensitivity to any components of the study drug, comparable drugs, or to latex.
9. Renal impairment: creatinine clearance <30 mL/min at screening or receiving dialysis.
10. Medical evidence of current or history of primary or secondary immunodeficiency.
11. Infection-related exclusions as further defined in the protocol.
12. Major surgical procedure within 8 weeks prior to the screening or scheduled during the study.
13. Current or history of any malignancy, or myeloproliferative, or lymphoproliferative disease within 5 years before screening.
14. History of clinically significant drug or alcohol abuse within the last year prior to randomization.
15. Prior denosumab (Prolia, Xgeva, or proposed denosumab biosimilar) exposure.
16. Prior use of fluoride within the 5 years before inclusion in the study.
17. Any current or prior use of strontium ranelate.
18. Any current or prior use of intravenous bisphosphonates.
19. Current or prior use of teriparatide and other parathormone (PTH) analogues within 12 months before screening.
20. Current or prior use of systemic oral or transdermal estrogen or selective estrogen receptor modulators or tibolone within 6 months before screening.
21. Current or prior use of calcitonin or cinacalcet within 3 months before screening or any cathepsin K inhibitor (eg, odanacatib) within 18 months before screening.
22. Current or prior use of romosozumab or antisclerostin antibody.
23. Current or prior use of other osteoporotic agents used for the prevention or treatment of osteoporosis.
24. Current use within 3 months before screening of any medication with known influence on the skeletal system (eg, systemic corticosteroids, heparin, lithium, etc) with exceptions described in the protocol.
25. Concomitant treatment with another biologic drug.
26. Have received a COVID-19 vaccine within 4 weeks before randomization or COVID-19 vaccination is ongoing at the time of screening.

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- Bulgaria (12):
  - Diagnostic Consultative Center Aleksandrovska, Sofia, Sofia-Grad
  - Diagnostic Consultative Center (DCC) 17 - Sofia, Sofia, Sofia-Grad
  - Medical Center N. I. Pirogov, Sofia, Sofia-Grad
  - Medical Center Hipokrat 2000 OOD, Haskovo
  - Medical Center Medconsult Pleven, Pleven
  - Palmed University Multidisciplinary Hospital for Active Treatment, Plovdiv
  - University Multi-profile Hospital for Active Treatment - Plovdiv, Plovdiv
  - Medical Center - Teodora EOOD, Rousse
  - Multiprofile Hospital for Active Treatment Hadzhi Dimitar, Sliven
  - Lyulin Hospital, Sofia
  - Diagnostic and Consultative Center Equita, Varna
  - Medical Center Sanador M, Vidin
- Czechia (6):
  - CCR Brno, Brno, Jihormoravsky Kraj
  - CCR Ostrava, Ostrava, Severomoravsky Kraj
  - Medical Plus, Uherské Hradiště, South Moravian
  - G-Centrum Olomouc s.r.o, Olomouc
  - Artroscan, Ostrava-T?ebovice
  - Medical Plus, Uherské Hradiště
- Estonia (5):
  - Center for Clinical and Basic Research AS - Tallinn, Tallinn, Harju
  - Sihtasutus Pohja-Eesti Regionaalhaigla, Tallinn, Harju
  - KLV Arstikabinet, Pärnu, Pärnumaa
  - Tartu Ulikooli Kliinikum, Tartu, Tartu
  - KLV Arstikabinet, Pärnu
- Georgia (7):
  - Evex Hospitals - Caraps Medline, Tbilisi, Borjomi
  - Georgian-Dutch Hospital, Tbilisi, Borjomi
  - Hepatology Clinic Hepa, Tbilisi
  - Tbilisi Heart And Vascular Clinic Ltd, Tbilisi
  - Jerarsi Clinic, Tbilisi
  - Raymann - Clinic of Raymann Doctors, Tbilisi
  - MedCity Ltd., Tbilisi
- Hungary (17):
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Szeged, Csongr
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Szeged, Csongrád megye
  - Csongrad-Csanad Megyei Dr. Bugyi Istvan Korhaz, Szentes, Csongrád megye
  - Szent Anna Magan N?gyogyaszati, Debrecen, Hajdú-Bihar
  - Markhot Ferenc Oktatokorhaz es Rendel?intezet, Eger, Heves County
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa, Pest County
  - Obudai Egeszsegugyi Centrum, Zalaegerszeg, Zala County
  - Drug Research Center Balatonfured, Balatonfüred
  - Revita Rendel?, Budapest
  - Clinexpert Gyogycentrum, Budapest
  - Obudai Egeszsegugyi Centrum, Budapest
  - Semmelweis Egyetem - I. sz. Belgyogyaszati Klinika, Budapest
  - Debreceni Egyetem Klinikai Kozpont Kenezy Gyula Campus, Debrecen
  - Markhot Ferenc Oktatokorhaz es Rendel?intezet, Eger
  - Kalocsai Szent Kereszt Korhaz, Kalocsa
  - CMed Rehabilitacios es Diagnosztikai Kozpont / Saldinvest Kft., Székesfehérvár
  - Vital Medical Center - Reumatologia, Veszprém
- Poland (28):
  - Centrum Medyczne Solumed, Pozna?, Greater Poland Voivodeship
  - Centrum Bada? Klinicznych, Poznan, Greater Poland Voivodeship
  - Nasz Lekarz Przychodnie Medyczne, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne All-Med, Krakow, Lesser Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - FutureMeds, Wroclaw, Lower Silesian Voivodeship
  - Wromedica Centrum Zdrowia, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Oporow, Wroclaw, Lower Silesian Voivodeship
  - RCMed Oddzial Sochaczew, Sochaczew, Masovian Voivodeship
  - Medycyna Kliniczna, Warsaw, Masovian Voivodeship
  - Centrum Medyczne AMED - Warszawa Targowek, Warsaw, Masovian Voivodeship
  - Rheuma Medicus - Specjalistyczne Centrum Reumatologii i Osteoporozy, Warsaw, Masovian Voivodeship
  - Twoja Przychodnia Szczeci?skie Centrum Medyczne, Warsaw, Masovian Voivodeship
  - SOMED CR - ?od?, Warsaw, Masovian Voivodeship
  - Osteo-Medic sc dr diabetolog Katarzyna Wasilewska, Bialystok, Podlaskie Voivodeship
  - ClinicMed, Bialystok, Podlaskie Voivodeship
  - Nasz Lekarz O?rodek Bada? Klinicznych - Bydgoszcz, Bydgoszcz, Pomeranian Voivodeship
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela w Bydgoszczy, Bydgoszcz, Pomeranian Voivodeship
  - Centrum Medyczne Pratia - Gdynia, Gdynia, Pomeranian Voivodeship
  - Gabinet diagnostyki i leczenia osteoporozy, Gliwice, Silesian Voivodeship
  - Centrum Kliniczno Badawcze J Brzezicki B Górnikiewicz Brzezicka Lekarze, Elblag, Warmian-Masurian Voivodeship
  - Ambulatorium Sp z o.o. - Elblag, Elblag, Zulawy
  - Centrum Medyczne All-Med, Krakow
  - SOMED CR - ?od?, Lodz
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Twoja Przychodnia Szczeci?skie Centrum Medyczne, Szczecin
  - Samodzielny Publiczny Zespo? Opieki Zdrowotnej w Tomaszow Lubelski, Tomaszów Lubelski
  - Klinika Reuma Park sp. z o.o. sp.k - Centrum Medyczne Reuma Park, Warsaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 553 participants were randomized in the study at 64 centers across 6 countries (Bulgaria, Czech Republic, Estonia, Georgia, Hungary, and Poland) between June 2021 and January 2022.
Pre-assignment Details: The study included a Screening Period of maximum 28 days prior to first drug (FKS518 and US-Prolia) administration, a double-blind Core Treatment Period up to Week 52, and a double-blind single Transition Period from Week 52 up to Week 78, with administration of the study drug on Day 1, Week 26, and Week 52.
Groups:
- Core Treatment Period FKS518: Participants received FKS518 60 mg subcutaneously on Day 1 and Week 26 during the Core Treatment Period (Baseline to Week 52).
- Core Treatment Period US-Prolia: Participants received US-Prolia 60 mg subcutaneously on Day 1 and Week 26 during the Core Treatment Period (Baseline to Week 52).
- Transition Period: FKS518 (Was on FKS518 in CTP): Participants treated with FKS518 during Core Treatment Period received FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
- Transition Period: FKS518 (Switched From US-Prolia in CTP): Participants treated with US-Prolia during Core period were re-randomised to receive FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
- Transition Period: US-Prolia (Was on US-Prolia in CTP): Participants treated with US-Prolia during Core period were continued to receive US-Prolia 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
Period: Day 0 to Week 52
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia | Transition Period: FKS518 (Was on FKS518 in CTP) | Transition Period: FKS518 (Switched From US-Prolia in CTP) | Transition Period: US-Prolia (Was on US-Prolia in CTP)
Started | 277 | 276 | 0 | 0 | 0
Completed (Re-randomized at Week 52) | 252 | 249 | 0 | 0 | 0
Not Completed | 25 | 27 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 22 | 0 | 0 | 0
Not completed — Discontinued Treatment Prior to Week 52 | 4 | 1 | 0 | 0 | 0
Not completed — Other | 3 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 0 | 0 | 0
Period: Week 52 to Week 78
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia | Transition Period: FKS518 (Was on FKS518 in CTP) | Transition Period: FKS518 (Switched From US-Prolia in CTP) | Transition Period: US-Prolia (Was on US-Prolia in CTP)
Started | 0 | 0 | 252 | 124 | 125
Completed | 0 | 0 | 245 | 122 | 122
Not Completed | 0 | 0 | 7 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 1 | 2
Not completed — Other | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) Analysis Set: The ITT Analysis Set included all randomized participants. Participants were analyzed according to their randomized treatment.
Groups:
- FKS518: FKS518: Participants received FKS518 60 mg subcutaneously on Day 1 and Week 26 during the Core Treatment Period (Baseline to Week 52).
- US-Prolia: US-Prolia: Participants received US-Prolia 60 mg subcutaneously on Day 1 and Week 26 during the Core Treatment Period (Baseline to Week 52).
- Total: Total of all reporting groups
Arm/Group | FKS518 | US-Prolia | Total
Number analyzed (Participants) | 277 | 276 | 553
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (6.44) | 65.8 (6.47) | 65.5 (6.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 276 | 553
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 277 | 276 | 553
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Lumbar spine bone mineral density (LS-BMD) by dual energy X-ray absorptiometry (DXA) [Mean (Standard Deviation); unit: g/cm^2] | 0.7872 (0.06381) | 0.7929 (0.05962) | 0.7901 (0.06176)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in LS-BMD by DXA
Description: Bone density was measured at the lumbar spine from L1 through L4. Per FDA request for this study, data were analyzed by non-inferiority and non-superiority analyses. Decreased BMD is associated with risk of fracture.
Time Frame: Baseline and Week 52
Population: ITT Analysis Set: The ITT Analysis Set included all randomized participants. Participants were analyzed according to their randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia
Number analyzed (Participants) | 277 | 276
Percentage change
  Non-Inferiority Analysis | 5.52 (0.292) | 5.07 (0.297)
  Non-Superiority Analysis | 5.73 (0.292) | 5.03 (0.297)
Statistical Analysis 1: Comparison: Core Treatment Period FKS518 vs Core Treatment Period US-Prolia; Test type: Non-Inferiority — Non-inferiority of FKS518 to US-Prolia was demonstrated if the 90% CI for the difference in mean percent change from baseline to Week 52 in LS-BMD laid entirely above -1.45%; Mean Difference (Final Values) = 0.46, 90% CI 2-sided [-0.05 to 0.96], Standard Error of Mean 0.306 — Difference : FKS518 - US-Prolia
Statistical Analysis 2: Comparison: Core Treatment Period FKS518 vs Core Treatment Period US-Prolia; Test type: Other — Non-superiority Analysis: Non-superiority of FKS518 to US-Prolia was demonstrated if the 90% CI for the difference in mean percent change from baseline to Week 52 in LS-BMD laid entirely below 1.45%; Mean Difference (Final Values) = 0.69, 90% CI 2-sided [0.19 to 1.20], Standard Error of Mean 0.306 — Difference : FKS518 - US-Prolia

2. Secondary Outcome: Area Under the Effect Curve (AUEC) of Serum C-terminal Cross-linking Telopeptide of Type 1 Collagen (CTX)
Description: Area under the effect curve for the (untransformed) biomarker concentrations from baseline up to Week 26. Any possible rebound effect where biomarker concentrations rose above baseline was not taken into account, and only the area below baseline was considered in this parameter.
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: (ng*h/L)
Groups:
- FKS518: Participants received FKS518 60 mg subcutaneously on Day 1 and Week 26 during the Core Treatment Period (Baseline to Week 52).
- US-Prolia: Participants received US-Prolia 60 mg subcutaneously on Day 1 and Week 26 during the Core Treatment Period (Baseline to Week 52).
Arm/Group | FKS518 | US-Prolia
Number analyzed (Participants) | 277 | 276
(ng*h/L) | 1884 [1840 to 1928] | 1862 [1818 to 1908]

3. Secondary Outcome: Percentage Change From Baseline in BMD at Femoral Neck and Total Hip by DXA
Description: The proximal femur (inclusive of femoral neck and total hip) DXA scans were obtained from the left side when possible. If the right side had to be used (e.g., due to implants) or was inadvertently used at baseline, then it had to be used consistently throughout the study. Data reported are for one half of the body only.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia
Number analyzed (Participants) | 277 | 276
Percentage change
  BMD at Femoral Neck at Week 52 | 2.07 (0.284) | 1.85 (0.291)
  BMD at Total Hip at Week 52 | 2.97 (0.217) | 2.88 (0.223)

4. Secondary Outcome: Percentage Change From Baseline in Serum Procollagen Type 1 N-terminal Propeptide (P1NP)
Description: P1NP is a bone biomarker. Serum samples were collected for analysis of P1NP to evaluate bone formation (P1NP) in response to treatment with FKS518 and US-Prolia. A decrease in the serum levels of P1NP is expected following treatment with denosumab and is suggestive of improvement.
Time Frame: Baseline and Week 52 pre dose
Population: Pharmacodynamic (PD) Analysis Set: All participants who received at least 1 dose of investigational product, had a quantifiable baseline PD marker concentration, and enough samples not impacted by protocol deviations to calculate the PD parameter. Only participants with available data are included.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia
Number analyzed (Participants) | 236 | 237
Percentage change | -65.27 (2.491) | -63.25 (2.536)

5. Secondary Outcome: Percentage Change From Baseline in Serum C-terminal Cross-linking Telopeptide of Type 1 Collagen (CTX)
Description: Serum CTX is a bone biomarker. Serum samples were collected for analysis of CTX to evaluate bone resorption in response to treatment with FKS518 or US-Prolia.
  A decrease in the serum levels of CTX is expected following treatment with US-Prolia and is suggestive of improvement.
Time Frame: Baseline and Week 52 pre dose
Population: PD Analysis Set: All participants who received at least 1 dose of investigational product, had a quantifiable baseline PD marker concentration, and enough samples not impacted by protocol deviations to calculate the PD parameter. Only participants with available data are included.
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia
Number analyzed (Participants) | 236 | 235
Percentage Change | -68.16 (4.241) | -64.47 (4.330)

6. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: Treatment-emergence was defined as AEs that began or increased in severity or frequency on or after the date of first administration of IP in a given treatment Period (Core or Transition) up to the Early Termination/End of Study Visit.
Time Frame: Day 1 to Week 78
Population: Safety Analysis Set (SAF): The SAF included all participants who received at least 1 dose of IP. The Transition Period Safety Analysis (TP-SAF) Set included all participants who received at least 1 dose of IP during the course of the TP. Participants were analyzed according to the actual treatment they received.
Measure: Count of Participants; unit: Participants
Groups:
- Core Treatment Period: FKS518; Transition Period: FKS518: Participants treated with FKS518 during Core Treatment Period received FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
- Core Treatment Period: US-Prolia; Transition Period: FKS518: Participants treated with US-Prolia during Core period were re-randomised to receive FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
- Core Treatment Period: US-Prolia; Transition Period: US-Prolia: Participants treated with US-Prolia during Core period were continued to receive US-Prolia 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
- Overall Period: FKS518: Participants treated with FKS518 during Core Treatment Period received FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78). This Reporting Group is used to report the results of the Overall period (Baseline to Week 78).
- Overall Period: Core Treatment Period: US-Prolia; Transition Period: FKS518: Participants treated with US-Prolia during Core period were re-randomised to receive FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78). This Reporting Group is used to report the results of the Overall period (Baseline to Week 78).
- Overall Period: US-Prolia: Participants treated with US-Prolia during Core period were continued to receive US-Prolia 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78). This Reporting Group is used to report the results of the Overall period (Baseline to Week 78).
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia | Core Treatment Period: FKS518; Transition Period: FKS518 | Core Treatment Period: US-Prolia; Transition Period: FKS518 | Core Treatment Period: US-Prolia; Transition Period: US-Prolia | Overall Period: FKS518 | Overall Period: Core Treatment Period: US-Prolia; Transition Period: FKS518 | Overall Period: US-Prolia
Number analyzed (Participants) | 277 | 276 | 252 | 124 | 125 | 277 | 124 | 152
Participants | 185 | 189 | 106 | 58 | 47 | 202 | 102 | 103

7. Secondary Outcome: Number of Participants Who Experienced a Treatment-Emergent Serious Adverse Event (TESAE)
Description: Treatment-emergence was defined as SAEs that began or increased in severity or frequency on or after the date of first administration of IP up to the Early Termination/End of Study Visit.
Time Frame: Day 1 to Week 78
Population: SAF: SAF included all participants who received at least 1 dose of IP. The TP-SAF Set included all participants who received at least 1 dose of IP during the course of the TP. Participants were analyzed according to the actual treatment they received.
Measure: Count of Participants; unit: Participants
Groups:
- Core Treatment Period: FKS518; Transition Period: FKS518: Participants treated with FKS518 during Core Treatment Period received FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78). This Reporting Group is used to report the results of the Transition period (Week 52 to 78).
- Core Treatment Period: US-Prolia; Transition Period: FKS518: Participants treated with US-Prolia during Core period were re-randomised to receive FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78). This Reporting Group is used to report the results of the Transition period (Week 52 to 78).
- Core Treatment Period: US-Prolia; Transition Period: US-Prolia: Participants treated with US-Prolia during Core period were continued to receive US-Prolia 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78). This Reporting Group is used to report the results of the Transition period (Week 52 to 78).
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia | Core Treatment Period: FKS518; Transition Period: FKS518 | Core Treatment Period: US-Prolia; Transition Period: FKS518 | Core Treatment Period: US-Prolia; Transition Period: US-Prolia | Overall Period: FKS518 | Overall Period: Core Treatment Period: US-Prolia; Transition Period: FKS518 | Overall Period: US-Prolia
Number analyzed (Participants) | 277 | 276 | 252 | 124 | 125 | 277 | 124 | 152
Participants | 43 | 50 | 8 | 6 | 6 | 50 | 27 | 33

8. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event of Special Interest (AESI)
Description: A Treatment-emergent AESI is defined as drug-related hypersensitivity/allergic reactions (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≥3 or reported as serious adverse events [SAEs]) and AEs leading to IP discontinuation or study withdrawal.
Time Frame: Day 1 to Week 78
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Core Treatment Period: US-Prolia; Transition Period: US-Prolia: Participants (125) treated with US-Prolia during Core period were continued to receive US-Prolia 60 mg subcutaneously, every 26 weeks during the Transition Period. This Reporting Group is used to report the results of the Transition period (Week 52 to 78).
- Overall Period: FKS518: Participants received FKS518 60 mg subcutaneously, every 26 weeks during the Core Treatment Period (Baseline to Week 52) and then continued to receive FKS518 treatment 60 mg subcutaneously, every 26 weeks during the Transition Period (Week 52 to Week 78). This Reporting Group is used to report the results of the Overall period (Baseline to Week 78).
- Overall Period: Core Treatment Period: US-Prolia; Transition Period: FKS518: Participants who were originally randomized to receive US-Prolia during core treatment period (Baseline to Week 52) were re-randomized to receive FKS518 subcutaneously; 60 mg every 26 weeks during transition treatment period (Week 52 to Week 78). This Reporting Group is used to report the results of the Overall period (Baseline to Week 78).
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia | Core Treatment Period: FKS518; Transition Period: FKS518 | Core Treatment Period: US-Prolia; Transition Period: FKS518 | Core Treatment Period: US-Prolia; Transition Period: US-Prolia | Overall Period: FKS518 | Overall Period: Core Treatment Period: US-Prolia; Transition Period: FKS518 | Overall Period: US-Prolia
Number analyzed (Participants) | 277 | 276 | 252 | 124 | 125 | 277 | 124 | 152
Participants | 0 | 7 | 0 | 1 | 0 | 0 | 1 | 7

9. Secondary Outcome: Number of Participants Who Experienced an Injection Site Reaction (ISR)
Description: Local tolerability in terms of ISRs was assessed by inspection of the skin and appendages in proximity to the site of administration. The injection site was the abdomen, and the IP was injected slowly. This local tolerability assessment was performed by the Investigator or designee to determine the presence of e.g., erythema, rash, tenderness, swelling, itching, bruising, pain, extravasation, phlebitis, or other types of reaction. The Investigator was also requested to ask participants during assessment about any such reactions that may have occurred since last assessment.
Time Frame: Day 1 to Week 78
Population: SAF: The SAF included all participants who received at least 1 dose of IP. The TP-SAF Set included all participants who received at least 1 dose of IP during the course of the TP. Participants were analyzed according to the actual treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Core Treatment Period FKS518 | Core Treatment Period US-Prolia | Core Treatment Period: FKS518; Transition Period: FKS518 | Core Treatment Period: US-Prolia; Transition Period: FKS518 | Core Treatment Period: US-Prolia; Transition Period: US-Prolia | Overall Period: FKS518 | Overall Period: Core Treatment Period: US-Prolia; Transition Period: FKS518 | Overall Period: US-Prolia
Number analyzed (Participants) | 277 | 276 | 252 | 124 | 125 | 277 | 124 | 152
Participants | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 78
Description: The SAF included all participants who received at least 1 dose of IP. All adverse events occurring in the Core Period and Transition Period are presented.
  Participants were analyzed according to the actual treatment they received.
Groups:
- Core Treatment Period: FKS518: Participants received FKS518 60 mg subcutaneously on Day 1 and Week 26 during the Core Treatment Period (Baseline to Week 52).
- Core Treatment Period: US-Prolia: Participants received US-Prolia 60 mg subcutaneously on Day 1 and Week 26 during the Core Treatment Period (Baseline to Week 52).
- Transition Treatment Period: FKS518 (Was on FKS518 in CTP): Participants treated with FKS518 during Core Treatment Period received FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
- Transition Treatment Period: US-Prolia (Was on US-Prolia in CTP): Participants treated with US-Prolia during Core period were continued to receive US-Prolia 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
- Transition Treatment Period: FKS518 (Switched From US-Prolia in CTP): Participants treated with US-Prolia during Core period were re-randomized to receive FKS518 60 mg subcutaneously on Week 52 during the Transition Period (Week 52 to Week 78).
Arm/Group | Core Treatment Period: FKS518 | Core Treatment Period: US-Prolia | Transition Treatment Period: FKS518 (Was on FKS518 in CTP) | Transition Treatment Period: US-Prolia (Was on US-Prolia in CTP) | Transition Treatment Period: FKS518 (Switched From US-Prolia in CTP)
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/276 | 0/252 | 0/125 | 0/124
Serious Adverse Events (participants affected / at risk) | 43/277 | 50/276 | 8/252 | 6/125 | 6/124
Other Adverse Events (participants affected / at risk) | 69/277 | 78/276 | 22/252 | 15/125 | 24/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Treatment Period: FKS518 (N=277) | Core Treatment Period: US-Prolia (N=276) | Transition Treatment Period: FKS518 (Was on FKS518 in CTP) (N=252) | Transition Treatment Period: US-Prolia (Was on US-Prolia in CTP) (N=125) | Transition Treatment Period: FKS518 (Switched From US-Prolia in CTP) (N=124)
COVID-19 (Infections and infestations) | 32 | 41 | 6 | 3 | 4
Asymptomatic COVID-19 (Infections and infestations) | 3 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Hydrometra (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Treatment Period: FKS518 (N=277) | Core Treatment Period: US-Prolia (N=276) | Transition Treatment Period: FKS518 (Was on FKS518 in CTP) (N=252) | Transition Treatment Period: US-Prolia (Was on US-Prolia in CTP) (N=125) | Transition Treatment Period: FKS518 (Switched From US-Prolia in CTP) (N=124)
Nasopharyngitis (Infections and infestations) | 26 (33) | 33 (41) | 11 (12) | 8 (8) | 17 (18)
Upper respiratory tract infection (Infections and infestations) | 23 (29) | 30 (36) | 12 (14) | 7 (7) | 8 (8)
Urinary tract infection (Infections and infestations) | 18 (22) | 23 (28) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (14) | 14 (15) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT04934072/Prot_SAP_000.pdf